CLINICAL TRIAL: NCT02915276
Title: Comparison of Genomic DNA Analysis Between Blastocoele Fluid and Trophectoderm Biopsy in Human Embryos
Brief Title: The Effectiveness of Blastocentesis Versus Trophectoderm Biopsy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Center for Reproductive an Genetic Health (Industry)
Responsible Party: Principal Investigator, Kalliopi Loutradi, Deputy Head of Embryology, Center for Reproductive an Genetic Health
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: blatocentesesJBNKL2016
Record Dates: First submitted 2016-09-22; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Abnormal Karyotype
Keywords: Blastocyst; Human; DNA; Blastocentesis
MeSH Terms: conditions — Abnormal Karyotype

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blastocentisis (Active Comparator): The blastocoelic fluid will be aspirated from the embryonic cavity on day 5 or 6 of development and will be subjected to genetic analysis
  Interventions: Procedure: Blastocentisis
- Trophectoderm biopsy (Active Comparator): Throphectoderm cells will be removed from the embryo on day 5 or 6 of development and will be subjected to genetic analysis
  Interventions: Procedure: Trophectoderm biopsy

INTERVENTIONS:
Procedure: Blastocentisis — Removal of blastocoelic fluid from the blastocoelic cavity
  Arms: Blastocentisis
Procedure: Trophectoderm biopsy — Removal of trophectoderm cells from the blastocyst
  Arms: Trophectoderm biopsy

SUMMARY:
For the purpose of this study, the investigators will perform the removal of trophectoderm (TE) the cells as required for the purpose of pre-implantation genetic screening, in order to perform the genetic analysis. Additionally, the investigators will remove the blastocoelic fluid (BF) and perform additional genetic analysis on the embryo in order to determine the agreement of the genetics results between TE cells and BF.

DETAILED DESCRIPTION:
The human embryo (fertilised egg) develops from a single cell and goes through several developmental stages in order to prepare for implantation inside the womb. During the fifth and sixth day post fertilisation, the embryo becomes a blastocyst. It consists of 100-150 cells and has two cell types. The inner cell mass (ICM) will give rise to the baby and the trophectoderm cells will become the placenta. The trophectoderm (TE) cells surround the ICM. Following the formation of the two cell types, the TE cells start producing fluid. The progressive accumulation of fluid leads to the formation of a cavity that expands to form the blastocele cavity. This cavity contains fluid is known as blastocoelic fluid (BF). The fluid can contain proteins, cells and genetic material. Traditionally to make a genetic diagnosis or when to screen embryos for abnormal chromosome number, cells are removed (biopsy) from the trophectoderm. In experienced hands, this is a very safe procedure and causes minimal damage to the embryo. However, recent studies have shown that blastocoele fluid may contain genetic material which can be aspirated (drawn out) from the blastocole cavity (blastocentesis) and used for genetic analysis of an embryo. This is potentially less invasive and harmful to the embryo. The aim of this study is to compare genetic analysis obtained following blastocentesis versus trophectoderm cell biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Couples undergoing assisted reproduction for pre-implantation genetic diagnosis

Exclusion Criteria:

* Any other couples undergoing assisted reproduction

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Number of blastocyst with genomic DNA present in the blastocoelic cavity | Twelve months

CONTACTS AND LOCATIONS:
Locations (1):
- Kalliopi Loutradi, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Magli MC, Pomante A, Cafueri G, Valerio M, Crippa A, Ferraretti AP, Gianaroli L. Preimplantation genetic testing: polar bodies, blastomeres, trophectoderm cells, or blastocoelic fluid? Fertil Steril. 2016 Mar;105(3):676-683.e5. doi: 10.1016/j.fertnstert.2015.11.018. Epub 2015 Dec 1. PMID 26658131
- [Result] Gianaroli L, Magli MC, Pomante A, Crivello AM, Cafueri G, Valerio M, Ferraretti AP. Blastocentesis: a source of DNA for preimplantation genetic testing. Results from a pilot study. Fertil Steril. 2014 Dec;102(6):1692-9.e6. doi: 10.1016/j.fertnstert.2014.08.021. Epub 2014 Sep 23. PMID 25256935